CLINICAL TRIAL: NCT04447261
Title: Safety, Tolerability, and Pharmacokinetics of Multiple Rising Oral Doses of BI 1356225 (Randomised, Placebo-controlled, Blinded Within Dose Groups) and Evaluation of Midazolam and Celecoxib Interaction (Nested, Open, Fixed-sequence, Intra-individual Comparison) in Patients With Overweight or Obesity
Brief Title: A Study to Test How Well Different Doses of BI 1356225 Are Tolerated by Men and Women With Obesity or Overweight
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: 1427-0002; 2020-000342-34 (EudraCT Number)
Record Dates: First submitted 2020-06-24; First posted 2020-06-25 (Actual); Last update posted 2021-05-19 (Actual); Status verified 2021-05

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- BI 1356225 (Experimental)
  Interventions: Drug: BI 1356225
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BI 1356225 — BI 1356225
  Arms: BI 1356225
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The primary objective of this trial is to investigate safety and tolerability of BI 1356225 in male and female patients with overweight and obesity following oral administration of multiple rising doses per day over 28 days. Secondary objectives are the exploration of pharmacokinetics (PK) of BI 1356225 after multiple oral dosing. Additionally, the relative bioavailability (BA) of midazolam and celecoxib in the presence and absence of BI 1356225 will be evaluated

ELIGIBILITY:
Inclusion criteria

* Male and female patients, age ≥ 18 and < 70
* Body Mass Index ≥ 27 kg/m2 and < 40 kg/m2 at screening
* Stable body weight (defined as no more than 5% change) within 3 months prior to screening
* further inclusion criteria apply

Exclusion criteria

* Females of childbearing potential
* Clinically relevant concomitant disease per investigator judgment
* Any condition or disease requiring permanent pharmacotherapy during the trial
* Any history of lifetime suicidal behaviour and any suicidal ideation of type 2 - 5 in the Columbia-Suicide Severity Rating Scale (C-SSRS) in the past 12 months
* further exclusion criteria apply

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2020-06-30 (Actual); Primary Completion 2021-04-25 (Actual); Study Completion 2021-04-25 (Actual)

PRIMARY OUTCOMES:
The percentage of subjects with drug-related adverse events | Up to 40 days

SECONDARY OUTCOMES:
AUCτ, 1 (area under the concentration-time curve of BI 1356225 in plasma over a uniform dosing interval τ after administration of the first dose) | Up to 35 days
Cmax,1 (maximum measured concentration of BI 1356225 in plasma after administration of the first dose) | Up to 35 days
AUCτ,ss (area under the concentration-time curve of BI 1356225 in plasma at steady state over a uniform dosing interval τ after administration of the last dose) | Up to 35 days
Cmax,ss (maximum measured concentration of BI 1356225 in plasma at steady state over a uniform dosing interval τ after administration of the last dose) | Up to 35 days
AUC0-tz (area under the concentration-time curve of midazolam in plasma over the time interval from 0 to the last quantifiable data point) | Up to 35 days
AUC0-tz (area under the concentration-time curve of celecoxib in plasma over the time interval from 0 to the last quantifiable data point) | Up to 35 days
Cmax (maximum measured concentration of midazolam in plasma) | Up to 35 days
Cmax (maximum measured concentration of celecoxib in plasma) | Up to 35 days

CONTACTS AND LOCATIONS:
Locations (1):
- CRS Clinical Research Services Mannheim GmbH, Mannheim, Germany

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents, except for the following exclusions: 1. studies in products where Boehringer Ingelheim is not the license holder; 2. studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; 3. studies conducted in a single center or targeting rare diseases (because of limitations with anonymization).For more details refer to: http://trials.boehringer-ingelheim.com/

REFERENCES:
- See also: Related Info — https://www.mystudywindow.com